CLINICAL TRIAL: NCT02391532
Title: Effect of Probiotic Bacteria (L. Reuteri) on Oral Candida Counts in Frail Elderly
Brief Title: Effect of Probiotic Bacteria on Oral Candida in Frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Rose Jørgensen, PhD Student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010/618
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri DSM 17938/ATCC PTA (Active Comparator): L. reuteri DSM 17938/ATCC PTA lozenges twice daily for 12 weeks
  Interventions: Dietary Supplement: L. reuteri DSM 17938/ATCC PTA
- Placebo (Placebo Comparator): Placebo lozenges twice daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938/ATCC PTA — Ingestion of active lozenge twice daily for 12 weeks
  Arms: L. reuteri DSM 17938/ATCC PTA
Dietary Supplement: Placebo — Ingestion of placebo lozenge twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of daily intake of the probiotic Lactobacillus Reuteri on the prevalence and counts of oral Candida in frail elderly living in nursery homes.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the effect of a twice daily intake of lozenges containing probiotic Lactobacillus reuteri on the prevalence and counts of oral Candida in senior residents living in nursery homes. The material consists of 215 elderly persons (range 60 to 102 years) living in 20 different nursery homes in the County of Kronoberg, situated in the southern parts of Sweden. The subjects were consecutively enrolled after informed consent consisting of verbal and written information directed to the individual as well as to their relatives. The study employed a double-blind randomized placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* ability to cooperate with a dental examination and saliva sampling

Exclusion Criteria:

* severe chronic disease, malignancies or ongoing medication with immunosuppressive drugs
* severe dementia or cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of oral Candida growth assessed from chair-side tests. | Baseline and 12 weeks.
  Saliva and plaque samples will be analyzed and data presented when all 215 participants have completed the intervention period.
Amount of oral Candida growth assessed from chair-side tests. | Baseline and 12 weeks.
  Saliva and plaque samples will be analyzed and data presented when all 215 participants have completed the intervention period.

SECONDARY OUTCOMES:
Change in levels of dental plaque | Baseline and 12 weeks.
  Secondary Outcome Measures will be measured before and after the intervention period.
Changes in levels of gingival bleeding. | Baseline and 12 weeks.
  Secondary Outcome Measures will be measured before and after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Svante Twetman, Professor, Study Director — University of Copenhagen

REFERENCES:
- [Derived] Kraft-Bodi E, Jorgensen MR, Keller MK, Kragelund C, Twetman S. Effect of Probiotic Bacteria on Oral Candida in Frail Elderly. J Dent Res. 2015 Sep;94(9 Suppl):181S-6S. doi: 10.1177/0022034515595950. Epub 2015 Jul 22. PMID 26202995